CLINICAL TRIAL: NCT06328803
Title: A Randomized Controlled Trial to Explore The Effect of Active Breathing Exercises in Stroke Patients With Respiratory Rhythm Disorder
Brief Title: Impact of Active Breathing Exercises on Respiratory Rhythm Disorders in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copka Sonpashan (Other Government)
Responsible Party: Sponsor-Investigator, Copka Sonpashan, The Research Director, Chao Phya Abhaibhubejhr Hospital
Organization: Chao Phya Abhaibhubejhr Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Active Breathing Exercises
Record Dates: First submitted 2024-03-10; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation training+Active Breathing Exercises (Experimental): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Based on this, this group was given Active Breathing Exercises
  Interventions: Behavioral: Rehabilitation training; Behavioral: Active Breathing Exercises
- Rehabilitation training (Active Comparator): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  Interventions: Behavioral: Rehabilitation training

INTERVENTIONS:
Behavioral: Rehabilitation training — Including 1) Basic treatment, including corresponding control of risk factors and education on healthy lifestyles. 2)Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
Behavioral: Active Breathing Exercises — Active breathing exercises aim to enhance the strength and flexibility of respiratory muscles through a series of exercises, improving breathing patterns and increasing respiratory efficiency. The following are common components of active breathing exercises: 1) Deep Breathing. 2) Chest Expansion. 3) Diaphragmatic Breathing. 4) Coughing Techniques. 5) Expiratory Resistance Training. 6) Gradual Increase in Activity.
  Arms: Rehabilitation training+Active Breathing Exercises

SUMMARY:
The goal of this clinical trial is to explore The Effect of Active Breathing Exercises in Stroke Patients With Respiratory Rhythm Disorder. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will be given Active Breathing Exercises. Researchers will compare dysphagia of two groups.

DETAILED DESCRIPTION:
A growing body of literature indicates the existence of a highly stable, coordinative relation between respiration and oropharyngeal swallowing in healthy adults. The goal of this clinical trial is to explore The Effect of Active Breathing Exercises in Stroke Patients With Respiratory Rhythm Disorder. Patients will be randomly divided into an observation group and a control group, all receiving routine rehabilitation treatment. On this basis, the observation group will be given Active Breathing Exercises. Researchers will compare dysphagia of two groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Respiratory Rhythm Disorder
* age ≥ 18 years;
* meeting the diagnostic criteria of stroke;
* any degree of dysphagia at admission;
* steady vital signs, without severe cognitive impairment or sensory aphasia, able to cooperate with the assessment.
* transferred out within three weeks of hospitalization in the neurology department.

Exclusion Criteria:

* complicated with other neurological diseases;
* tracheostomy tube plugged;
* unfeasible to the support of parenteral nutrition;
* simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 15
  The Penetration-Aspiration Scale is used to assess the severity of airway invasion during swallowing. The score ranges from 1 to 8, with higher scores indicating more severe penetration or aspiration events. A lower score indicates better swallowing function and less risk of airway invasion, while a higher score suggests more significant impairment and increased risk of aspiration.

SECONDARY OUTCOMES:
Functional Oral Intake Scale | day 1 and day 15
  The Functional Oral Intake Scale is used to measure the level of oral intake and diet consistency in individuals with dysphagia. The score ranges from 1 to 7, with higher scores indicating better functional oral intake and tolerance to a wider variety of food textures. A higher score indicates improved swallowing function and the ability to consume a better range of food consistencies, while a lower score suggests more significant impairments and a limited intake of oral food and liquids.
Yale Pharyngeal Residue Severity Rating Scale | day 1 and day 15
  The Yale Pharyngeal Residue Severity Rating Scale is used to assess the severity of pharyngeal residue after swallowing. The scale ranges from 1 to 5, with higher scores indicating worse severity of pharyngeal residue. A higher score on the Yale Pharyngeal Residue Severity Rating Scale indicates a larger amount of residue remaining in the pharynx after swallowing, while a lower score suggests less residue and better swallowing efficiency.
Fiberoptic Endoscopic Dysphagia Severity Scale | day 1 and day 15
  The Fiberoptic Endoscopic Dysphagia Severity Scale is used to assess the severity of swallowing disorders based on fiberoptic endoscopic examination. The score ranges from 1 to 8, with higher scores indicating more severe swallowing impairment.
Murray Secretion Scale | day 1 and day 15
  The Murray Secretion Scale is used to assess the amount and tenacity of tracheobronchial secretions. The score ranges from 0 to 4, with higher scores indicating a greater amount and/or thicker consistency of secretions. A higher score indicates a higher volume or thicker consistency of tracheobronchial secretions, while a lower score suggests minimal secretion accumulation and easier secretion management.
Swallowing Quality of Life | day 1 and day 15
  Swallowing Quality of Life is a self-report questionnaire designed to assess the impact of dysphagia on an individual's quality of life. The score ranges from 0 to 100, with higher scores indicating better swallowing-related quality of life. A higher score indicates a better quality of life related to swallowing function, while a lower score suggests a poorer quality of life and greater negative impact of dysphagia on daily activities and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group